CLINICAL TRIAL: NCT01680107
Title: The Effect of a Single-dose of D-cycloserine on the Basic Effects of Cognitive-behaviour Therapy for Panic Disorder - a Randomized Placebo-controlled Trial
Brief Title: D-cycloserine Augmented CBT for Panic Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MRC-01; 2012-003191-39 (EudraCT Number)
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Panic Disorder
Keywords: d-cycloserine, cognitive-behaviour therapy, panic disorder
MeSH Terms: conditions — Panic Disorder | interventions — Cycloserine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- d-cycloserine (Experimental): oral, capsule, 250 mg, once
  Interventions: Drug: d-cycloserine; Behavioral: cognitive-behaviour therapy
- sugar pill (Placebo Comparator): oral, capsule, once
  Interventions: Drug: placebo; Behavioral: cognitive-behaviour therapy

INTERVENTIONS:
Drug: d-cycloserine
  Arms: d-cycloserine
Drug: placebo
  Arms: sugar pill
Behavioral: cognitive-behaviour therapy

SUMMARY:
The purpose of this study is to determine whether d-cycloserine augments the clinical effects of exposure-based cognitive-behaviour therapy for panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of panic disorder
* at least moderate agoraphobic avoidance

Exclusion Criteria:

* psychoactive medication last 6 weeks
* exposure-based cognitive-behaviour treatment for panic disorder and agoraphobia during last 3 months
* female participant who is pregnant or breast-feeding
* lifetime history of psychosis, bipolar disorder, alcohol, medication or drug abuse or dependence; current primary depressive disorder
* lifetime history of epilepsy or other significant disease or disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2017-10-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
self-reported and clinician-rated anxiety and depression measures | 6 months

SECONDARY OUTCOMES:
emotional information processing | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Reinecke, PhD, Principal Investigator — University of Oxford; Catherine Harmer, PhD, Study Director — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Reinecke A, Nickless A, Browning M, Harmer CJ. Neurocognitive processes in d-cycloserine augmented single-session exposure therapy for anxiety: A randomized placebo-controlled trial. Behav Res Ther. 2020 Jun;129:103607. doi: 10.1016/j.brat.2020.103607. Epub 2020 Mar 19. PMID 32229324